CLINICAL TRIAL: NCT04497870
Title: Peppermint Oil Pharmacokinetics/Dynamics and Novel Biological Signatures in Children With Functional Abdominal Pain
Brief Title: Peppermint Oil Pharmacokinetics/Dynamics
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was superseded by NCT03295747
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Shulman, M.D., Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-40351
Record Dates: First submitted 2020-06-22; First posted 2020-08-04 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — peppermint oil; Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 540 mg (Active Comparator): Peppermint oil at a dose of 180 mg thrice daily orally
  Interventions: Drug: Peppermint oil
- 900 mg (Experimental): Peppermint oil at a dose of 180 mg five times daily orally
  Interventions: Drug: Peppermint oil

INTERVENTIONS:
Drug: Peppermint oil — Administration of peppermint oil at one of two daily doses.
  Other Names: menthol

SUMMARY:
In children 7-12 years of age with functional abdominal pain (n=42) determine:

Aim 1 - To examine and characterize the threshold of the exposure (PK) vs. response (PD) relationship of PMO (menthol)

Aim 2 - PD of PMO as assessed by:

1. Microbiome composition (16S RNA sequencing)
2. Transit rate/contractile activity (using the SmartPill®) Aim 3 - Evaluate the potential association between PD response and clinical symptoms (abdominal pain and stooling pattern via validated diary), psychosocial distress (anxiety, depression, somatization), and characterize potential side effects (questionnaire)

DETAILED DESCRIPTION:
An initial single-dose PK study will be carried out. Forty-two children (n=21 per dose) will be randomized to receive approximately 10.9 mg·kg-1·d-1 of PMO or to receive approximately 18.2 mg·kg-1·d-1 (1.67-fold the median dose).

Following the single-dose PK study, a PD study will be carried out wherein the subjects will receive their assigned dose of PMO for 7 days.

At baseline (before the PK study) and after the PK study (i.e., during the PD study), subjects will keep a pain and stooling diary, collect stool for microbiome analysis, and swallow a SmartPill to measure gut motility and transit time. At baseline only, anxiety, depression, somatization will be measured. During the PD study, any side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-12 years who are able to assent to the procedures
* Able to complete the diaries which have been validated for use in this age range
* The history and medical evaluation reveal no organic reason for the abdominal pain
* The child has abdominal pain that meets the definition of FAP according to pediatric Rome IV
* Ability to understand study procedures and to comply with them for the entire length of the study
* Childrens' body weights will not vary by more than 10-15 kg (so that dose per kg is comparable within the two dosing groups)

Exclusion Criteria:

* Past bowel surgery
* Documented GI disorders (e.g., Crohn's disease)
* A serious chronic medical condition (e.g., diabetes)
* A weight and/or height < 2 SD for age
* Chronic conditions with GI symptoms (e.g., cystic fibrosis)
* Autism spectrum disorder, significant developmental delay, psychosis, depression, or a history of bipolar disorder
* Antibiotic/probiotic treatment within 2 mo.
* Allergy/sensitivity to PMO or its ingredients
* Inability to swallow the PMO capsule or the SmartPill®
* Inability to speak English - testing materials are available only in this language
* Unable to discontinue laxative, prokinetic, or neuromodulator from 3 wk prior to Visit 1 through the end of the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of peppermint oil | 2 weeks
  Area under the curve
Gut Microbiome composition | 2 weeks
  Gut microbiome composition as determined by 16S sequencing as a consequence of the administration of peppermint oil at the two doses given.
Gut transit time | 2 weeks
  Gut transit time as a consequence of the administration of peppermint oil at the two doses given.
Gut contractility | 2 weeks
  Gut contractility as a consequence of the administration of peppermint oil at the two doses given.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Shulman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No